CLINICAL TRIAL: NCT02884297
Title: Feasibility Study of the Measurement of the Placental Perfusion During the First Trimester of Pregnancy by 3D Doppler Echo-angiography With a Contrast Agent
Brief Title: HexafluOride, a Contrast Agent for Placenta Echo-angiography
Acronym: HOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-01-CHRMT
Record Dates: First submitted 2016-07-14; First posted 2016-08-31 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy
MeSH Terms: interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgical termination of pregnancy (Experimental): Contrast agent: SonoVue®: Hexafluoride (SonoVue®, injectable solution to solubilisate, 8µg/mL) is injected in all patients for ultrasound angiography during the termination of pregnancy. 2,4 mL are administrated per patient, divided into two injections of 1,2 mL.
  Interventions: Drug: Contrast agent: SonoVue®.

INTERVENTIONS:
Drug: Contrast agent: SonoVue®. — SonoVue® Injection: will be done through the peripheral venous way already set up by the anesthetist for its injection. None venous dedicated way will be established. The injection will take place when the woman will be under general anesthesia, ventilated and under constant cardio-respiratory monitoring.
  Other Names: hexafluoride

SUMMARY:
The purpose of this study is to quantify the placental perfusion during the first trimester of pregnancy by 3D Doppler ultrasound angiography without a contrast agent and by ultrasound with a contrast agent: SonoVue®

DETAILED DESCRIPTION:
The quality of the utero-placental vascularization is a major point for the foetal healthy development and for the healthy pregnancy. Pre-eclampsia (PE) and the Intra-Uterine Growth Retardation (IUGR) are currently two of the major pregnancy complications in the West. Those placental pathologies cause more than 30 per cent of the foetal and maternal morbidity-mortality. The relationship between these pathologies, affecting 4 to 7 per cent of pregnancies, and a chronic utero-placental hypoperfusion, which is caused by a failure of implantation during the first trimester of pregnancy, has been confirmed.

A hypoxic environment surrounds the embryonic implantation and the first steps of the placental development into uterus. Moreover, the maternal-foetal exchanges space (the Inter-Villi Space or IVS) is so maternal-bloodless. At the pregnancy first period are released there uterine secretions and a plasmatic ultra-filtrate. Indeed, the ends of the uterine arteries are plugged by trophoblastic plugs.

It was also accepted that the disappearance of these plugs, a major step in the implementation of the mother-fetal interface, occurred around 10 weeks of amenorrhea (10 SA). However, a recent study questions this dogma since the presence of blood in the intervilleous chamber has just been detected as early as 6 weeks of amenorrhea (6SA). In addition, an increase in blood flow within the IVS is found between 6 and 13 SA. Thus, it would appear that chronic placental hypoperfusion phenomena are more related to a vascular flow defect within the IVS than to the disappearance of endovascular plugs.

These new advances come from a single recent publication which was carried out on a small number of people (maximum 4 women per group).

It is therefore essential to carry out further studies to confirm that the infusion of IVS occurs very early and to evaluate the evolution of infusion kinetics with gestational age.

The detection of blood in the IVS from 6 SA was made possible by the injection of an ultrasound vascular contrast agent. This contrast agent does not have marketing authorization in women and its use is therefore not possible during the course of the progressive desired pregnancies. This study can therefore only be conducted in women who have confirmed a desire for voluntary interruption of pregnancy.

Since 2004, the quantification of the placental and uterine vascularization is possible by Doppler 3D ultrasound angiography but this technique has only been evaluated from 11SA. The advantage of this technique is that it does not require the injection of contrast agent, but the main limitation is that the Doppler signal observed is not necessarily specific to a blood flow. Thus, it would be interesting to evaluate whether 3D Doppler ultrasound angiography would make it possible to quantify the perfusion of the IVS early, compared to contrast ultrasound. If this is the case, the use of contrast media would no longer be necessary to evaluate the evolution of placental flux in future studies.

Recent data challenge ideas that have been accepted for decades. It is crucial to continue early exploration in order to understand the kinetics of maternal blood development in the IVS.

This kinetic would have a major impact on the progression of pregnancy and it analysis may permit a screening test and an early diagnosis for PE- or IUGR-risky pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and <65 years,
* Gestational Age: 8 SA ≤ gestational age ≤ 8 SA + 6 days or 11 SA ≤ gestational age ≤ 11 SA + 6 days,
* BMI ≤40 kg / m²,
* Having confirmed his request for termination of pregnancy surgically

Exclusion Criteria:

1. Any medical contraindication for administration of

   SonoVue including:
   * Hypersensitivity to sulfur hexafluoride or any of the other components of SonoVue®,
   * Women with recent acute coronary syndrome or suffering from an unstable ischemic heart disease,
   * women having a right-left shunt, severe pulmonary hypertension (pulmonary artery pressure> 90 mmHg), an uncontrolled systemic hypertension and woman with respiratory distress syndrome
2. Women with risk for IUGR / PE namely:

   * Previous history of PE or stunting staff
   * Autoimmune disease,
   * Chronic Hypertension
   * Diabetes

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The measurement of signal strength | 1 day
  The measurement of signal strength (in arbitrary units) in the Inter-Villi Space in the first trimester (at 8SA, 11SA and 13SA) obtained by contrast ultrasound, in women who have confirmed a voluntary termination of pregnancy.

SECONDARY OUTCOMES:
Measurement of the vascularization parameters of the Inter-Villi Space (IVS) and myometrium: signal strength | 1 day
  Measurement of the vascularization parameters of the Inter-Villi Space (IVS) and myometrium: signal strength
Measurement of the vascularization parameters of the Inter-Villi Space (IVS) and myometrium: infusion kinetics. | 1 day
  Measurement of the vascularization parameters of the Inter-Villi Space (IVS) and myometrium: infusion kinetics.
Comparison of quantitative data on uteroplacental vascularization obtained with the 2 techniques. | 1 day
  Comparison of quantitative data on uteroplacental vascularization obtained with the 2 techniques: by 3D Doppler ultrasound angiography without a contrast agent and by ultrasound with a contrast agent: SonoVue®.
Obtaining analyzable placental villi for the study of the development and functions of the human placenta. | 1 day
  Obtaining analyzable placental villi for the study of the development and functions of the human placenta.
  Placental tissue collected will be analyzed to better understand the development and function of the placenta during pregnancy in a subsequent search. The genetic polymorphism research of some placental genes may also be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure ESZTO-CAMBON, MD, Principal Investigator — CHR Metz-Thionville
Locations (2):
- France (2):
  - Chr Metz Thionville, Metz
  - CHRU de NANCY, Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bertholdt C, Eszto ML, Tournier M, Hossu G, Mellouki N, Cherifi A, Morel O. Assessment of uteroplacental vascularisation in early first-trimester pregnancy with contrast-enhanced ultrasound and 3D power Doppler angiography: protocol for a prospective, cross-sectional, multicentre and non-randomised open study ("HOPE Study"). BMJ Open. 2019 Sep 11;9(9):e030353. doi: 10.1136/bmjopen-2019-030353. PMID 31511289